CLINICAL TRIAL: NCT00103285
Title: Standard Risk B-precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Combination Chemotherapy in Treating Young Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL0331; NCI-2009-00302 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 05-340; COG-AALL0331; CDR0000409589; AALL0331 (Other: Children's Oncology Group); AALL0331 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia; Childhood B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Radiotherapy, Conformal; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Thioguanine; Vincristine

ARMS (8):
- Group 0 Induction Therapy (Experimental): All patients receive cytarabine intrathecally (IT) on day 1; vincristine IV on days 1, 8, 15, and 22; dexamethasone IV or orally (PO) twice daily (BID) on days 1-28; pegaspargase intramuscularly (IM) (may give IV over 1 to 2 hours) on day 4, 5, or 6; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease). Patients with Down syndrome (DS) receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT. Patients are assessed for response on day 29. Patients with M1 bone marrow AND minimal residual disease (MRD) < 0.1% OR MRD >= 0.1% and < 1% proceed to therapy in part II. Patients with M2 bone marrow OR M1 bone marrow AND MRD >= 1% proceed to extended induction therapy. Patients with M3 bone marrow are removed from the study.
  Interventions: Drug: Cytarabine; Drug: Dexamethasone; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine Sulfate
- Group 1-SR-low ALL, Arm I (combination chemotherapy) (Active Comparator): Patients receive standard consolidation therapy, standard interim maintenance therapy, and standard delayed intensification (DI) therapy, followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group 1-SR-low ALL, arm II (combination chemotherapy) (Experimental): Patients receive experimental consolidation therapy, experimental interim maintenance therapy, and standard DI therapy, followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Dexamethasone; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine Sulfate
- Group 2-SR-avg ALL, arm I (combination chemotherapy) (Active Comparator): Patients receive standard consolidation therapy, standard interim maintenance therapy, and standard DI therapy as in group 1, arm I, followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine
- Group 2-SR-avg ALL, arm II (combination chemotherapy) (Experimental): Patients receive standard consolidation therapy, augmented interim maintenance therapy, augmented DI therapy, followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group 2-SR-avg ALL, arm III (combination chemotherapy) (Active Comparator): Patients receive intensified consolidation therapy, standard interim maintenance therapy, and standard DI therapy, followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group 2-SR-avg ALL, arm IV (combination chemotherapy) (Active Comparator): Patients receive intensified consolidation therapy, augmented interim maintenance therapy, and augmented DI therapy, followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Group 3-SR-high ALL, combination chemotherapy (Experimental): Patients receive intensified consolidation therapy, augmented interim maintenance therapy (2 courses), and augmented DI therapy (2 courses), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Some patients undergo cranial radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
  Arms: Group 1-SR-low ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm I (combination chemotherapy); Group 2-SR-avg ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Group 1-SR-low ALL, Arm I (combination chemotherapy); Group 2-SR-avg ALL, arm I (combination chemotherapy); Group 2-SR-avg ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy
Drug: Cytarabine — Given IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Group 0 Induction Therapy; Group 1-SR-low ALL, Arm I (combination chemotherapy); Group 2-SR-avg ALL, arm I (combination chemotherapy); Group 2-SR-avg ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV or IT
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Group 1-SR-low ALL, Arm I (combination chemotherapy); Group 2-SR-avg ALL, arm I (combination chemotherapy); Group 2-SR-avg ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy
Drug: Leucovorin Calcium — Given PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Group 1-SR-low ALL, Arm I (combination chemotherapy); Group 1-SR-low ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm I (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy
Drug: Methotrexate — Given IM or IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Group 1-SR-low ALL, Arm I (combination chemotherapy); Group 2-SR-avg ALL, arm I (combination chemotherapy); Group 2-SR-avg ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Group 0 Induction Therapy; Group 1-SR-low ALL, Arm I (combination chemotherapy); Group 1-SR-low ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm II (combination chemotherapy); Group 2-SR-avg ALL, arm III (combination chemotherapy); Group 2-SR-avg ALL, arm IV (combination chemotherapy); Group 3-SR-high ALL, combination chemotherapy

SUMMARY:
This randomized phase III trial is studying different combination chemotherapy regimens and comparing how well they work in treating patients with newly diagnosed acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the substitution of three intensified phases of post-Induction treatment for standard phases will improve the event free survival (EFS) of children with SR-average acute lymphoblastic leukemia (ALL).

II. Determine whether the substitution of intensified Consolidation for standard Consolidation will improve the EFS of children with SR-average ALL.

III. To determine whether the addition of four doses of percutaneous endoscopic gastrostomy (PEG) asparaginase, given once every three weeks during Consolidation and Interim Maintenance phases, will improve the EFS for children with SR-low ALL.

SECONDARY OBJECTIVES:

I. Identify potentially modifiable factors associated with impaired health related quality of life (HRQOL) at different periods of therapy in the patients who are SR-average enrolled on the standard risk ALL study.

II. Determine the critical time periods when future intervention studies to mitigate adverse HRQOL outcomes should occur.

III. Correlate day 29 minimal residual disease (MRD) with EFS and overall survival (OS) of patients treated with these regimens.

IV. Correlate early marrow response with day 29 MRD status. V. To improve outcome by identifying additional high risk patients by Day 29 MRD for treatment with fully augmented Berlin-Frankfurt-Munster (BFM).

VI. To examine the relative contributions of genetic factors and early treatment response to outcome by comparing the outcome of patients with and without TEL-AML1 fusion or triple trisomy and low levels of MRD at end Induction who are treated with identical therapy on the standard arms of the SR-low and SR-average trials.

OUTLINE: This is a 2-part, partially randomized, multicenter study. Patients are stratified according to early response to study induction therapy (rapid early response [standard risk (SR)-low or SR-average acute lymphoblastic leukemia (ALL)] vs slow early response [SR-high ALL]). After completion of induction therapy but before proceeding to part II therapy, patients are assigned to 1 of 3 groups based on stratification.

PART I:

INDUCTION THERAPY: All patients receive cytarabine intrathecally (IT) on day 1; vincristine IV on days 1, 8, 15, and 22; dexamethasone IV or orally (PO) twice daily (BID) on days 1-28; pegaspargase intramuscularly (IM) (may give IV over 1 to 2 hours) on day 4, 5, or 6; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease). Patients with Down syndrome (DS) receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT. Patients are assessed for response on day 29. Patients with M1 bone marrow AND minimal residual disease (MRD) < 0.1% OR MRD >= 0.1% and < 1% proceed to therapy in part II. Patients with M2 bone marrow OR M1 bone marrow AND MRD >= 1% proceed to extended induction therapy. Patients with M3 bone marrow are removed from the study.

EXTENDED INDUCTION THERAPY: Patients receive dexamethasone IV or PO BID on days 1-14; vincristine IV on days 1 and 8; pegaspargase IM on day 4, 5, or 6; and daunorubicin hydrochloride IV over 15 minutes to 2 hours on day 1. Patients with M1 bone marrow and MRD < 1% after extended induction therapy proceed to therapy in part II. Patients with M2 or M3 bone marrow after extended induction therapy are removed from the study.

PART II:

GROUP 1 (SR-low ALL): Patients are randomized to 1 of 2 treatment arms.

ARM I:

STANDARD CONSOLIDATION THERAPY: Patients receive vincristine IV on day 1; mercaptopurine PO on days 1-28; and methotrexate IT on days 1, 8, and 15. Patients with Down syndrome (DS) receive leucovorin calcium (PO) at 48 and 60 hours after each dose of methotrexate IT.

STANDARD INTERIM MAINTENANCE THERAPY: Patients receive vincristine IV on days 1 and 29; dexamethasone IV or PO BID on days 1-5 and 29-33; mercaptopurine PO on days 1-50; methotrexate PO on days 1, 8, 15, 22, 29, 36, 43, and 50; and methotrexate IT on day 29. Patients with DS receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT.

STANDARD DELAYED INTENSIFICATION (DI) THERAPY: Patients receive vincristine IV on days 1, 8, and 15; dexamethasone IV or PO BID on days 1-21; doxorubicin hydrochloride IV over 15 minutes to 2 hours on days 1, 8, and 15; pegaspargase IM on day 4, 5, or 6; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV or subcutaneously (SC) on days 29-32 and 36-39; thioguanine PO on days 29-42; and methotrexate IT on days 1 and 29. Patients with DS receive dexamethasone IV or PO BID on days 1-7 and 15-21 and leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT.

ARM II:

EXPERIMENTAL CONSOLIDATION THERAPY: Patients receive vincristine, mercaptopurine, methotrexate, and leucovorin calcium as in arm I and pegaspargase IM on days 1 and 22.

EXPERIMENTAL INTERIM MAINTENANCE THERAPY: Patients receive vincristine, dexamethasone, mercaptopurine, methotrexate PO, and methotrexate IT as in arm I and pegaspargase IM on days 15 and 36.Standard DI therapy: Patients receive standard DI therapy as in arm I.

GROUP 2 (SR-average ALL): Patients are randomized to 1 of 4 treatment arms.

ARM I: Patients receive standard consolidation therapy, standard interim maintenance therapy, and standard DI therapy as in group 1, arm I.

ARM II:

STANDARD CONSOLIDATION THERAPY: Patients receive standard consolidation therapy as in group 1, arm I. Augmented interim maintenance therapy: Patients receive vincristine IV and methotrexate IV on days 1, 11, 21, 31, and 41; pegaspargase IM on days 2 and 22; and methotrexate IT on days 1 and 31. Patients with DS receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT. Augmented DI therapy: Patients receive vincristine IV on days 1, 8, 15, 43, and 50; dexamethasone IV or PO BID on days 1-21; doxorubicin hydrochloride IV over 15 minutes to 2 hours on days 1, 8, and 15; pegaspargase IM on day 4, 5, or 6 AND day 43; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV or SC on days 29-32 and 36-39; thioguanine PO on days 29-42; and methotrexate IT on days 1, 29, and 36. Patients with DS receive dexamethasone on days 1-7 and 15-21 and leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT.

ARM III:

INTENSIFIED CONSOLIDATION THERAPY: Patients receive cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine IV or SC on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO on days 1-14 and 29-42; vincristine IV on days 15, 22, 43, and 50; pegaspargase IM on days 15 and 43; and methotrexate IT on days 1, 8, 15*, and 22*. Patients with DS receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT*.

NOTE: *Patients with CNS3 disease at diagnosis do not receive methotrexate on days 15 and 22 or leucovorin calcium.

STANDARD INTERIM MAINTENANCE THERAPY: Patients receive standard interim maintenance therapy as in group 1, arm I.

STANDARD DI THERAPY: Patients receive standard DI therapy as in group 1, arm I.

ARM IV:

INTENSIFIED CONSOLIDATION THERAPY: Patients receive intensified consolidation therapy as in group 2, arm III.

AUGMENTED INTERIM MAINTENANCE THERAPY: Patients receive augmented interim maintenance therapy as in group 2, arm II.

AUGMENTED DI THERAPY: Patients receive augmented DI therapy as in group 2, arm II.

GROUP 3 (SR-high ALL): Patients receive the following therapy: Intensified consolidation therapy: Patients receive intensified consolidation therapy as in group 2, arm III.

AUGMENTED INTERIM MAINTENANCE* THERAPY: Patients receive augmented interim maintenance therapy as in group 2, arm II. Treatment repeats every 56 days for 2 courses.

NOTE: *As of Amendment #7, all SR-High patients currently receiving AIM 1 therapy should complete this phase of therapy and proceed to ADI 1 therapy as originally planned including Capizzi methotrexate during AIM 1. Upon completion of ADI 1, patients should receive a second Interim Maintenance phase with high-dose methotrexate (IM HD) rather than Capizzi methotrexate. Patients should then proceed to ADI 2 and then Maintenance.

AUGMENTED DI* THERAPY: Patients receive augmented DI therapy as in group 2, arm II. Treatment repeats every 56 days for 2 courses**.

NOTE: *As of Amendment #7, all SR-High patients currently receiving ADI 1 therapy should complete this phase of therapy as originally planned. Upon completion of ADI 1, patients should receive a second Interim Maintenance phase with IM HD. Patients should then proceed to ADI 2 and then Maintenance.

NOTE: **Patients with CNS3 disease at diagnosis also undergo cranial radiotherapy on days 29-33 and 36-40 during course 2 only; these patients do not receive methotrexate on day 36, thioguanine, or leucovorin calcium.

MAINTENANCE THERAPY: All patients receive vincristine IV on days 1, 29, and 57; oral dexamethasone twice daily on days 1-5, 29-33, and 57-61; oral methotrexate on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; oral mercaptopurine on days 1-84; and methotrexate IT* on day 1. Courses repeat every 84 days for a total of 2 years from the start of interim maintenance therapy for female patients and 3 years from the start of interim maintenance therapy for male patients.

NOTE: *SR-High or CNS3 patients should receive up to a maximum of 23 intrathecal treatments for females and 26 intrathecal treatments for males.

After the completion of study treatment, patients are followed every 1-2 months for 2 years, every 3 months for 1 year, and then every 6-12 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on AALL03B1 prior to enrollment on AALL0331
* Initial white blood cells (WBC) < 50,000/ul
* Newly diagnosed B-precursor acute lymphoblastic leukemia

  * Standard-risk (SR) disease meeting 1 of the following criteria:
  * SR-average by age and WBC
  * No unfavorable features
  * Rapid early responder (RER) by day 15
  * CNS 1 or 2
  * Minimal residual disease (MRD) negative on day 29
  * Trisomies of 4, 10, and 17 or TEL-AML1 translocation and RER and CNS2 allowed
  * SR-low by age and WBC
  * No unfavorable features
  * RER by day 15
  * MRD negative on day 29
  * CNS1
  * Favorable cytogenetics-trisomies of 4, 10, and 17 or TEL-AML translocation
  * SR-high
  * Unfavorable features meeting ≥ 1 of the following criteria:

    * MLL rearrangements and RER
    * Steroid pretreatment
    * CNS3
    * Slow early responder by morphology or MRD
* Patients with Down syndrome are allowed
* Patients with overt testicular disease are not eligible for this study, but may be eligible for AALL0232
* Patients shall have had no prior cytotoxic chemotherapy with the exception of steroids and intrathecal cytarabine; intrathecal chemotherapy with cytarabine is allowed prior to registration for patient convenience; this is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture; (Note: the central nervous system [CNS] status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment
* Patients receiving prior steroid therapy may be eligible for AALL0331 study
* Patients with a contraindication to additional asparaginase therapy, following Induction, are not eligible for the Standard Risk-Low study, and should be removed from protocol therapy at the end of Induction
* Patients who are assigned to the standard risk-average group following Induction and who meet the HRQOL
* Age at diagnosis >= 2 years (note that this is a more restrictive age range than for the therapeutic component of the study)
* At least one parent with reading comprehension of English or Spanish languages for which validated surveys exist
* Diagnosis at one of the institutions participating in this limited institution correlative study
* A parent or legal guardian must sign a written informed consent/parental permission for all patients
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5377 (Actual)
Dates: Start 2005-04-11 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly W Maloney, Principal Investigator — Children's Oncology Group
Locations (236):
- United States (210):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Brookdale Hospital Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (3):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Children's Hospital, Wellington
- Switzerland (3):
  - Swiss Pediatric Oncology Group - Bern, Bern
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Derived] Chen W, Chang TC, Rabin KR, Raetz EA, Devidas M, Hunger SP, Ramirez NC, Mullighan CG, Loh ML, Wu G. Performance of Two-Phase Designs for the Time-to-Event Outcome and a Case Study Assessing the Relapse Risk Associated With B-ALL Subtypes. JCO Clin Cancer Inform. 2025 May;9:e2400223. doi: 10.1200/CCI-24-00223. Epub 2025 May 2. PMID 40315406
- [Derived] Chang TC, Chen W, Qu C, Cheng Z, Hedges D, Elsayed A, Pounds SB, Shago M, Rabin KR, Raetz EA, Devidas M, Cheng C, Angiolillo A, Baviskar P, Borowitz M, Burke MJ, Carroll A, Carroll WL, Chen IM, Harvey R, Heerema N, Iacobucci I, Wang JR, Jeha S, Larsen E, Mattano L, Maloney K, Pui CH, Ramirez NC, Salzer W, Willman C, Winick N, Wood B, Hunger SP, Wu G, Mullighan CG, Loh ML. Genomic Determinants of Outcome in Acute Lymphoblastic Leukemia. J Clin Oncol. 2024 Oct 10;42(29):3491-3503. doi: 10.1200/JCO.23.02238. Epub 2024 Aug 9. PMID 39121442
- [Derived] Escherich CS, Chen W, Li Y, Yang W, Nishii R, Li Z, Raetz EA, Devidas M, Wu G, Nichols KE, Inaba H, Pui CH, Jeha S, Camitta BM, Larsen E, Hunger SP, Loh ML, Yang JJ. Germ line genetic NBN variation and predisposition to B-cell acute lymphoblastic leukemia in children. Blood. 2024 May 30;143(22):2270-2283. doi: 10.1182/blood.2023023336. PMID 38446568
- [Derived] Rabin KR, Devidas M, Chen Z, Ji L, Kairalla J, Hitzler JK, Yang JJ, Carroll AJ, Heerema NA, Borowitz MJ, Wood BL, Roberts KG, Mullighan CG, Harvey RC, Chen IM, Willman CL, Reshmi SC, Gastier-Foster JM, Bhojwani D, Rheingold SR, Maloney KW, Mattano LA, Larsen EC, Schore RJ, Burke MJ, Salzer WL, Winick NJ, Carroll WL, Raetz EA, Loh ML, Hunger SP, Angiolillo AL. Outcomes in Children, Adolescents, and Young Adults With Down Syndrome and ALL: A Report From the Children's Oncology Group. J Clin Oncol. 2024 Jan 10;42(2):218-227. doi: 10.1200/JCO.23.00389. Epub 2023 Oct 27. PMID 37890117
- [Derived] Wood B, Wu D, Crossley B, Dai Y, Williamson D, Gawad C, Borowitz MJ, Devidas M, Maloney KW, Larsen E, Winick N, Raetz E, Carroll WL, Hunger SP, Loh ML, Robins H, Kirsch I. Measurable residual disease detection by high-throughput sequencing improves risk stratification for pediatric B-ALL. Blood. 2018 Mar 22;131(12):1350-1359. doi: 10.1182/blood-2017-09-806521. Epub 2017 Dec 28. PMID 29284596
- [Derived] Karol SE, Mattano LA Jr, Yang W, Maloney KW, Smith C, Liu C, Ramsey LB, Fernandez CA, Chang TY, Neale G, Cheng C, Mardis E, Fulton R, Scheet P, San Lucas FA, Larsen EC, Loh ML, Raetz EA, Hunger SP, Devidas M, Relling MV. Genetic risk factors for the development of osteonecrosis in children under age 10 treated for acute lymphoblastic leukemia. Blood. 2016 Feb 4;127(5):558-64. doi: 10.1182/blood-2015-10-673848. Epub 2015 Nov 20. PMID 26590194
- [Derived] Teachey DT, Rheingold SR, Maude SL, Zugmaier G, Barrett DM, Seif AE, Nichols KE, Suppa EK, Kalos M, Berg RA, Fitzgerald JC, Aplenc R, Gore L, Grupp SA. Cytokine release syndrome after blinatumomab treatment related to abnormal macrophage activation and ameliorated with cytokine-directed therapy. Blood. 2013 Jun 27;121(26):5154-7. doi: 10.1182/blood-2013-02-485623. Epub 2013 May 15. PMID 23678006
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1-SR-low ALL, Arm I-combination Chemotherapy; Group 2-SR-avg ALL, Arm I-combination Chemotherapy: Patients receive standard consolidation therapy (vincristine sulfate, mercaptopurine and methotrexate. Patients with Down syndrome (DS) receive leucovorin calcium), standard interim maintenance therapy (vincristine sulfate, dexamethasone, mercaptopurine and methotrexate. Patients with DS receive leucovorin calcium), and standard delayed intensification (DI) therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine and methotrexate. Patients with DS receive dexamethasone, leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
- Group 1-SR-low ALL, Arm II-combination Chemotherapy: Patients receive experimental consolidation therapy (vincristine sulfate, mercaptopurine, MTX, leucovorin calcium and pegaspargase), experimental interim maintenance therapy (vincristine sulfate, dexamethasone, mercaptopurine, MTX and pegaspargase), and standard DI therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine and MTX), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
- Group 2-SR-avg ALL, Arm II-combination Chemotherapy: Patients receive standard consolidation therapy (vincristine sulfate, mercaptopurine and MTX. Patients with Down syndrome (DS) receive leucovorin calcium), augmented interim maintenance therapy (vincristine sulfate, MTX and pegaspargase. Patients with DS receive leucovorin calcium), augmented DI therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine, MTX. Patients with DS receive dexamethasone and leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
- Group 2-SR-avg ALL, Arm III-combination Chemotherapy: Patients receive intensified consolidation therapy (cyclophosphamide, cytarabine, mercaptopurine and vincristine sulfate, pegaspargase, MTX. Patients with DS receive oral leucovorin calcium), standard interim maintenance therapy (vincristine sulfate, dexamethasone, mercaptopurine and MTX. Patients with DS receive leucovorin calcium), and standard DI therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine and MTX. Patients with DS receive dexamethasone, leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
- Group 2-SR-avg ALL, Arm IV-combination Chemotherapy: Patients receive intensified consolidation therapy (cyclophosphamide, cytarabine, mercaptopurine and vincristine sulfate, pegaspargase, MTX. Patients with DS receive oral leucovorin calcium), augmented interim maintenance therapy (vincristine sulfate, MTX and pegaspargase. Patients with DS receive leucovorin calcium), and augmented DI therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine, MTX. Patients with DS receive dexamethasone and leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
- Group 3-SR-high ALL, Combination Chemotherapy: Patients receive intensified consolidation therapy (cyclophosphamide, cytarabine, mercaptopurine & vincristine sulfate, pegaspargase, methotrexate. Patients with DS receive oral leucovorin calcium), augmented interim maintenance therapy (2 courses - vincristine sulfate, methotrexate and pegaspargase. Patients with DS receive leucovorin calcium), and augmented DI therapy (2 courses - vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine, methotrexate. Patients with DS receive dexamethasone and leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  3-dimensional conformal radiation therapy: Some patients undergo cranial radiotherapy
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine
Period: Induction
Arm/Group | Group 0 Induction Therapy | Group 1-SR-low ALL, Arm I-combination Chemotherapy | Group 1-SR-low ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm I-combination Chemotherapy | Group 2-SR-avg ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm III-combination Chemotherapy | Group 2-SR-avg ALL, Arm IV-combination Chemotherapy | Group 3-SR-high ALL, Combination Chemotherapy
Started | 5377 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4028 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1349 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 103 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal | 906 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 258 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Response Assignment
Arm/Group | Group 0 Induction Therapy | Group 1-SR-low ALL, Arm I-combination Chemotherapy | Group 1-SR-low ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm I-combination Chemotherapy | Group 2-SR-avg ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm III-combination Chemotherapy | Group 2-SR-avg ALL, Arm IV-combination Chemotherapy | Group 3-SR-high ALL, Combination Chemotherapy
Started | 0 | 939 | 937 | 503 | 509 | 249 | 248 | 643
Completed | 0 | 807 | 853 | 441 | 425 | 201 | 199 | 523
Not Completed | 0 | 132 | 84 | 62 | 84 | 48 | 49 | 120
Not completed — Adverse Event | 0 | 8 | 3 | 2 | 3 | 1 | 1 | 2
Not completed — Death | 0 | 5 | 2 | 2 | 3 | 1 | 0 | 8
Not completed — Lost to Follow-up | 0 | 9 | 5 | 5 | 1 | 2 | 2 | 5
Not completed — Physician Decision | 0 | 13 | 14 | 9 | 13 | 7 | 4 | 35
Not completed — Protocol Violation | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 1 | 2 | 2 | 0 | 2
Not completed — Ineligible | 0 | 8 | 6 | 2 | 0 | 3 | 1 | 5
Not completed — Refusal | 0 | 53 | 5 | 3 | 25 | 15 | 30 | 10
Not completed — Other | 0 | 30 | 48 | 38 | 37 | 17 | 11 | 53

BASELINE CHARACTERISTICS:
Arm/Group | Group 0 Induction Therapy
Number analyzed (Participants) | 5377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5377
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.45 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2489
  Male | 2888
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1097
  Not Hispanic or Latino | 4038
  Unknown or Not Reported | 242
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 36
  Asian | 253
  Native Hawaiian or Other Pacific Islander | 24
  Black or African American | 326
  White | 4046
  More than one race | 0
  Unknown or Not Reported | 692
Region of Enrollment [Number; unit: participants]
  United States | 5377

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) for SR-Average ALL Patients
Description: EFS for SR-Average with standard and Intensified Consolidation. Event Free Probability where EFS time is defined as time from randomization to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free.
Time Frame: 6 years
Population: Only eligible patients are included in this population. Populations are based on enrollments for all four arms initially, and then only for Arms I and II (standard therapy) once Arms III and IV (intensified therapy) were closed to accrual.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Group 2-SR-avg ALL, Arm I-combination Chemotherapy | Group 2-SR-avg ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm III-combination Chemotherapy | Group 2-SR-avg ALL, Arm IV-combination Chemotherapy
Number analyzed (Participants) | 500 | 509 | 245 | 246
percent probability
  Standard and Intensified therapy: number analyzed (Participants) | 244 | 249 | 245 | 246
  Standard and Intensified therapy | 83.82 [78.86 to 88.78] | 88.89 [84.79 to 92.99] | 88.34 [83.99 to 92.69] | 90.51 [86.55 to 94.47]
  Standard therapy: number analyzed (Participants) | 500 | 509 | 0 | 0
  Standard therapy | 87.41 [83.63 to 91.19] | 88.29 [84.76 to 91.82] |  |

2. Primary Outcome: Event-free Survival (EFS) for SR-Low Patients
Description: Event Free Probability where EFS time is defined as time from randomization to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free.
Time Frame: 6 years
Population: Only eligible patients are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percent probability
Groups:
- SR-low ALL, Arm I-combination Chemotherapy: Patients receive standard consolidation therapy (vincristine sulfate, mercaptopurine and methotrexate. Patients with Down syndrome (DS) receive leucovorin calcium), standard interim maintenance therapy (vincristine sulfate, dexamethasone, mercaptopurine and methotrexate. Patients with DS receive leucovorin calcium), and standard delayed intensification (DI) therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine and methotrexate. Patients with DS receive dexamethasone, leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
- SR-low ALL, Arm II-combination Chemotherapy: Patients receive experimental consolidation therapy (vincristine sulfate, mercaptopurine, MTX, leucovorin calcium and pegaspargase), experimental interim maintenance therapy (vincristine sulfate, dexamethasone, mercaptopurine, MTX and pegaspargase), and standard DI therapy (vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine and MTX), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
  cyclophosphamide: Given IV
  thioguanine: Given PO
  vincristine sulfate: Given IV
Arm/Group | SR-low ALL, Arm I-combination Chemotherapy | SR-low ALL, Arm II-combination Chemotherapy
Number analyzed (Participants) | 928 | 929
Percent probability | 95.22 [93.6 to 96.9] | 93.96 [92.1 to 95.8]

3. Secondary Outcome: Health-related Quality of Life Relative to Physical, Social and Emotional Impairment
Description: To identify potentially modifiable factors associated with impaired health related quality of life (HRQOL) at different periods of therapy in the patients who are SR-average enrolled on the standard risk ALL study.Standardized scores will be computed for child function using the gender and age-adjusted scores available from normative data from a healthy population of about 10,000 children. The various domains of family functioning will be assessed using well-validated instruments and analyzed as a dichotomous variable (impaired vs. non-impaired family functioning). Multiple regression analysis will be used to test the effect of family functioning (adjusted for therapy given, age at diagnosis, gender, socioeconomic status and other factors) on child function.
Time Frame: At 1, 6 and 12 months after diagnosis and, 3 months post-therapy
Population: This analysis is restricted to the 160 SR-ALL patients enrolled on Children's Oncology Group (COG) therapeutic trial AALL0331 at 31 sites, who consented to and completed the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales (physical, emotional and social functioning).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Induction Therapy: All patients for induction therapy.
Arm/Group | Induction Therapy
Number analyzed (Participants) | 160
Percentage of participants
  Physical Impairment 1 mth after diagnosis | 76.39 [68.6 to 83.1]
  Physical Impairment 6 mths after diagnosis | 42.75 [34.2 to 51.7]
  Physical Impairment 12 mths after diagnosis | 29.41 [21.9 to 37.8]
  Physical Impairment 3 mths post therapy | 27.84 [19.2 to 37.9]
  Social Impairment 1 mth after diagnosis | 43.36 [35.1 to 51.9]
  Social Impairment 6 mths after diagnosis | 23.66 [16.7 to 31.9]
  Social Impairment 12 mths after diagnosis | 23.53 [16.7 to 31.6]
  Social Impairment 3 mths post-therapy | 25.77 [17.4 to 35.7]
  Emotional Impairment 1 mth after diagnosis | 38.89 [30.9 to 47.4]
  Emotional Impairment 6 mths after diagnosis | 17.56 [11.5 to 25.2]
  Emotional Impairment 12 mths after diagnosis | 13.97 [8.6 to 21.0]
  Emotional Impairment 3 mths post-therapy | 8.25 [3.6 to 15.6]
Statistical Analysis 1: Comparison: Induction Therapy; Physical Functioning: Parents of 160 SR-ALL patients enrolled on Children's Oncology Group (COG) therapeutic trial AALL0331 at 31 sites completed the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales (physical, emotional and social functioning) and Family Assessment Device-General Functioning (FAD-GF) at 1, 6 and 12 months after diagnosis, and 3 months post-therapy; Test type: Superiority or Other; Mixed Models Analysis; Odds Ratio (OR) = 5.17, 95% CI 2-sided [1.61 to 16.63] — Odds Ratios in this Statistical Analysis corresponds to all four time points
Statistical Analysis 2: Comparison: Induction Therapy; Social Functioning: Parents of 160 SR-ALL patients enrolled on Children's Oncology Group (COG) therapeutic trial AALL0331 at 31 sites completed the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales (physical, emotional and social functioning) and Family Assessment Device-General Functioning (FAD-GF) at 1, 6 and 12 months after diagnosis, and 3 months post-therapy; Test type: Superiority or Other; Mixed Models Analysis; Odds Ratio (OR) = 1.99, 95% CI 2-sided [1.21 to 3.27] — Odds Ratios in this Statistical Analysis corresponds to all four time points
Statistical Analysis 3: Comparison: Induction Therapy; Parents of 160 SR-ALL patients enrolled on Children's Oncology Group (COG) therapeutic trial AALL0331 at 31 sites completed the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales (physical, emotional and social functioning) and Family Assessment Device-General Functioning (FAD-GF) at 1, 6 and 12 months after diagnosis, and 3 months post-therapy; Test type: Superiority or Other; Mixed Models Analysis; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.03 to 3.34] — Odds Ratios in this Statistical Analysis corresponds to all four time points

4. Secondary Outcome: Event-Free Survival Probability According to MRD Status End Induction (Day 29)
Description: Event-Free survival by Day 29 MRD status (negative vs positive), Event Free Probability (time from study entry to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free.
Time Frame: MRD at Day 29 of therapy
Population: 4981 eligible evaluable patients enrolled on AALL0331 had MRD data at Day 29
Measure: Number (95% Confidence Interval); unit: Percent Probability
Groups:
- Induction Therapy, MRD Negative; Induction Therapy, MRD Positive: All patients receive cytarabine intrathecally (IT) on day 1; vincristine IV on days 1, 8, 15, and 22; dexamethasone IV or orally (PO) twice daily (BID) on days 1-28; pegaspargase intramuscularly (IM) (may give IV over 1 to 2 hours) on day 4, 5, or 6; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease). Patients with Down syndrome (DS) receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT. Patients are assessed for response on day 29. Patients with M1 bone marrow AND minimal residual disease (MRD) < 0.1% OR MRD >= 0.1% and < 1% proceed to therapy in part II. Patients with M2 bone marrow OR M1 bone marrow AND MRD >= 1% proceed to extended induction therapy. Patients with M3 bone marrow are removed from the study.
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  vincristine sulfate: Given IV
Arm/Group | Induction Therapy, MRD Negative | Induction Therapy, MRD Positive
Number analyzed (Participants) | 4614 | 367
Percent Probability | 91.39 [90.41 to 92.37] | 79.86 [75.04 to 84.68]
Statistical Analysis 1: Comparison: Induction Therapy, MRD Negative vs Induction Therapy, MRD Positive; 4981 eligible evaluable patients enrolled on AALL0331 had MRD evaluation at Day 29 of induction. MRD status defined as negative (<0.1%) or positive (>=0.1%). MRD status ( positive vs. negative) was correlated with EFS using Cox regression analysis; Test type: Superiority or Other; Regression, Cox; Hazard Ratio (HR) = 2.542, 95% CI 2-sided [1.974 to 3.273]

5. Secondary Outcome: Overall Survival Probability (OS) According to Induction Day 29 MRD Status
Description: Overall survival by Day 29 MRD status (negative vs positive), Overall survival defined as time from study entry to death or date of last contact for patients who are alive.
Time Frame: Overall Survival Probability of 6 years
Population: 4981 eligible evaluable patients enrolled on AALL0331 had MRD data at Day 29.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Induction Therapy, MRD Negative | Induction Therapy, MRD Positive
Number analyzed (Participants) | 4614 | 367
percent probability | 97.07 [96.5 to 97.68] | 90.47 [86.92 to 94.02]

6. Secondary Outcome: Early Marrow Status (EMS) by MRD Status End Induction (Day 29)
Description: Early Marrow Status defined as M1 versus M2/M3 marrow is correlated with MRD (Positive vs. Negative)
Time Frame: Early Marrow Status at Day 15, MRD Status at Day 29 of therapy.
Population: Patients who had MRD day 29 data but their Bone Marrow (BM) days 8/15 data were missing are excluded. This analysis was done with patients who had both MRD and BM data. There were 5 patients excluded in both MRD Negative and MRD Positive groups due to missing days 8/15 BM.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients for Induction, MRD Negative; All Patients for Induction, MRD Positive: All patients receive cytarabine intrathecally (IT) on day 1; vincristine IV on days 1, 8, 15, and 22; dexamethasone IV or orally (PO) twice daily (BID) on days 1-28; pegaspargase intramuscularly (IM) (may give IV over 1 to 2 hours) on day 4, 5, or 6; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease). Patients with Down syndrome (DS) receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT. Patients are assessed for response on day 29. Patients with M1 bone marrow AND minimal residual disease (MRD) < 0.1% OR MRD >= 0.1% and < 1% proceed to therapy in part II. Patients with M2 bone marrow OR M1 bone marrow AND MRD >= 1% proceed to extended induction therapy. Patients with M3 bone marrow are removed from the study.
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  vincristine sulfate: Given IV
Arm/Group | All Patients for Induction, MRD Negative | All Patients for Induction, MRD Positive
Number analyzed (Participants) | 4609 | 362
Participants | 4378 | 258
Statistical Analysis 1: Comparison: All Patients for Induction, MRD Negative vs All Patients for Induction, MRD Positive; MRD status ( positive vs. negative) was correlated with Early Marrow Status (M1 vs M2/M3) using Chi Square test; Test type: Superiority or Other; Chi-squared; Odds Ratio (OR) = 0.131, 95% CI 2-sided [0.101 to 0.17]

7. Secondary Outcome: Optimal Time Point for Advance Health Related Quality of Life Intervention
Description: Percentage of patients with elevated Anxiety.
Time Frame: At 1 month after diagnosis and 3 months post-therapy.
Population: Parents of 159 SR-ALL patients enrolled on Children's Oncology Group (COG) therapeutic trial AALL0331 at 31 sites completed the BASC-2 Anxiety Scale at 1 month after diagnosis, and 3 months post-therapy. Of these, 159 patients had data at 1 month after diagnosis and 96 patients had data at 3 months post therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Induction Therapy: All patients receive cytarabine intrathecally (IT) on day 1; vincristine IV on days 1, 8, 15, and 22; dexamethasone IV or orally (PO) twice daily (BID) on days 1-28; pegaspargase intramuscularly (IM) (may give IV over 1 to 2 hours) on day 4, 5, or 6; and methotrexate IT on days 8 and 29 (and days 15 and 22 for patients with CNS3 disease). Patients with Down syndrome (DS) receive leucovorin calcium PO at 48 and 60 hours after each dose of methotrexate IT. Patients are assessed for response on day 29. Patients with M1 bone marrow AND minimal residual disease (MRD) < 0.1% OR MRD >= 0.1% and < 1% proceed to therapy in part II. Patients with M2 bone marrow OR M1 bone marrow AND MRD >= 1% proceed to extended induction therapy. Patients with M3 bone marrow are removed from the study.
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  vincristine sulfate: Given IV
Arm/Group | Induction Therapy
Number analyzed (Participants) | 159
Percentage of participants
  At 1 month after diagnosis | 25.2 [18.5 to 31.9]
  At 3 months post-therapy: number analyzed (Participants) | 96
  At 3 months post-therapy | 24.0 [16.0 to 32.0]
Statistical Analysis 1: Comparison: Induction Therapy; Parents of 159 SR-ALL patients enrolled on Children's Oncology Group (COG) therapeutic trial AALL0331 at 31 sites completed the BASC-2 Anxiety Scale at 1 month after diagnosis, and 3 months post-therapy. Of these 159 had data at 1 month after diagnosis and 96 at 3 months post therapy; Test type: Other; Regression, Logistic; Odds Ratio (OR) = 4.1, 95% CI 2-sided [1.31 to 12.73]

8. Secondary Outcome: Event-free Survival (EFS) for SR-High Patients.
Description: as for outcome 2
Time Frame: 6 years
Population: CCR: Complete Continuous Remission, where time to event is defined as the time from start of consolidation therapy to first event or date of last follow up for those who did not experience an event. All patients enrolled on the SR-High were used in this analysis regardless of completion of therapy.
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- Group 3-SR-high ALL, Combination Chemotherapy: Patients receive intensified consolidation therapy (cyclophosphamide, cytarabine, mercaptopurine and vincristine sulfate, pegaspargase, methotrexate. Patients with DS receive oral leucovorin calcium), augmented interim maintenance therapy (2 courses - vincristine sulfate, MTX and pegaspargase. Patients with DS receive leucovorin calcium, and augmented DI therapy (2 courses - vincristine sulfate, dexamethasone, doxorubicin hydrochloride, pegaspargase, cyclophosphamide, cytarabine, thioguanine,MTX. Patients with DS receive (dexamethasone and leucovorin calcium), followed by maintenance therapy. Therapies are given by mouth, injection, and infusion for up to 2 or 3 years.
  doxorubicin hydrochloride: Given IV or IT
  3-dimensional conformal radiation therapy: Some patients undergo cranial radiotherapy
  cytarabine: Given IV or SC
  dexamethasone: Given IV or PO
  pegaspargase: Given IM
  methotrexate: Given IM or IT
  leucovorin calcium: Given PO
  mercaptopurine: Given PO
Arm/Group | Group 3-SR-high ALL, Combination Chemotherapy
Number analyzed (Participants) | 636
percent probability | 85.58 [85.55 to 85.61]

9. Secondary Outcome: Event-Free Survival (EFS) for Low MRD (Negative) Subjects by Genetic Subset (TEL/Trisomy Positive vs Negative)
Description: Event-free probability where EFS is defined as time from randomization to first event (relapse, second malignant neoplasm, death) or date of last contact for patients who are event-free.
Time Frame: 6 years
Population: Patients on the two arms being compared got similar therapy. All patients included in this analysis are MRD negative. SR-Average patients who were CNS2 at diagnosis were excluded in order to have comparable patient cohorts. SR-Low patients are TEL/Trisomy positive while SR-Average patients are TEL/Trisomy negative.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Group 1-SR-low ALL, Arm I-combination Chemotherapy | Group 2-SR-avg ALL, Arm I-combination Chemotherapy
Number analyzed (Participants) | 926 | 422
Percent probability | 95.22 [93.58 to 96.86] | 88.52 [84.56 to 92.48]

ADVERSE EVENTS:
Description: Only eligible patients are included in the toxicity analysis.
Arm/Group | Group 0 Induction Therapy | Group 1-SR-low ALL, Arm I-combination Chemotherapy | Group 1-SR-low ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm I-combination Chemotherapy | Group 2-SR-avg ALL, Arm II-combination Chemotherapy | Group 2-SR-avg ALL, Arm III-combination Chemotherapy | Group 2-SR-avg ALL, Arm IV-combination Chemotherapy | Group 3-SR-high ALL, Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 29/1306 | 14/931 | 7/931 | 4/501 | 3/509 | 0/246 | 1/247 | 12/638
Other Adverse Events (participants affected / at risk) | 790/1306 | 901/931 | 909/931 | 487/501 | 500/509 | 237/246 | 234/247 | 629/638
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 0 Induction Therapy (N=1306) | Group 1-SR-low ALL, Arm I-combination Chemotherapy (N=931) | Group 1-SR-low ALL, Arm II-combination Chemotherapy (N=931) | Group 2-SR-avg ALL, Arm I-combination Chemotherapy (N=501) | Group 2-SR-avg ALL, Arm II-combination Chemotherapy (N=509) | Group 2-SR-avg ALL, Arm III-combination Chemotherapy (N=246) | Group 2-SR-avg ALL, Arm IV-combination Chemotherapy (N=247) | Group 3-SR-high ALL, Combination Chemotherapy (N=638)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cecal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalomyelitis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 6 (6) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 0 Induction Therapy (N=1306) | Group 1-SR-low ALL, Arm I-combination Chemotherapy (N=931) | Group 1-SR-low ALL, Arm II-combination Chemotherapy (N=931) | Group 2-SR-avg ALL, Arm I-combination Chemotherapy (N=501) | Group 2-SR-avg ALL, Arm II-combination Chemotherapy (N=509) | Group 2-SR-avg ALL, Arm III-combination Chemotherapy (N=246) | Group 2-SR-avg ALL, Arm IV-combination Chemotherapy (N=247) | Group 3-SR-high ALL, Combination Chemotherapy (N=638)
Anemia (Blood and lymphatic system disorders) | 86 (88) | 258 (438) | 232 (356) | 119 (183) | 127 (213) | 55 (113) | 90 (150) | 213 (466)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2) | 8 (16) | 6 (8) | 1 (1) | 4 (5) | 2 (2) | 1 (1) | 9 (9)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 130 (131) | 531 (1045) | 555 (1045) | 272 (513) | 330 (733) | 144 (259) | 150 (316) | 475 (1260)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 2 (2) | 8 (8) | 6 (7) | 4 (4) | 2 (2) | 3 (8) | 5 (5) | 7 (14)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 10 (10) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 24 (24) | 32 (38) | 27 (32) | 27 (32) | 24 (29) | 7 (10) | 15 (19) | 36 (42)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Anal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cecal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (6) | 7 (7) | 5 (5) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 10 (12)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (12) | 15 (17) | 12 (12) | 8 (10) | 10 (11) | 2 (2) | 5 (5) | 14 (15)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 24 (24) | 82 (91) | 63 (67) | 47 (56) | 44 (49) | 17 (20) | 26 (28) | 68 (88)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 6 (6) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 7 (7) | 4 (4) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 9 (10)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 5 (5) | 2 (2) | 3 (3) | 5 (6)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 10 (10) | 8 (9) | 5 (5) | 3 (3) | 7 (7) | 2 (2) | 3 (3) | 4 (4)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 9 (9) | 62 (64) | 53 (61) | 36 (42) | 41 (52) | 19 (28) | 23 (28) | 81 (93)
Nausea (Gastrointestinal disorders) | 6 (6) | 14 (14) | 9 (10) | 14 (16) | 11 (12) | 2 (2) | 4 (4) | 21 (25)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3) | 11 (13) | 5 (5) | 14 (17) | 10 (12) | 3 (3) | 5 (5) | 18 (18)
Pancreatic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 18 (19) | 6 (7) | 2 (3) | 5 (6) | 9 (12) | 3 (3) | 5 (7) | 20 (28)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 6 (6) | 9 (9) | 6 (6) | 1 (1) | 8 (8) | 3 (3) | 3 (3) | 11 (13)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 11 (11) | 48 (53) | 37 (42) | 36 (47) | 33 (40) | 19 (24) | 18 (19) | 52 (65)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 16 (16) | 2 (2) | 8 (11) | 8 (9) | 3 (3) | 2 (2) | 11 (11)
Fever (General disorders) | 6 (6) | 84 (104) | 108 (128) | 49 (58) | 53 (66) | 36 (45) | 20 (23) | 71 (84)
Flu like symptoms (General disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 6 (6) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 5 (6) | 9 (13) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 7 (7)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 2 (3) | 6 (9) | 4 (6) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 5 (5)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 9 (9) | 14 (14) | 14 (14) | 2 (2) | 7 (8) | 8 (9) | 2 (2) | 19 (26)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 9 (10) | 4 (5) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 10 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 4 (4) | 76 (83) | 9 (9) | 5 (5) | 62 (66) | 31 (32) | 32 (35) | 92 (102)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 2 (2) | 2 (4) | 5 (5)
Abdominal infection (Infections and infestations) | 2 (2) | 8 (9) | 14 (14) | 4 (4) | 5 (6) | 5 (5) | 4 (4) | 6 (7)
Anorectal infection (Infections and infestations) | 0 (0) | 9 (9) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Appendicitis (Infections and infestations) | 2 (2) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arteritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 3 (3) | 10 (10) | 10 (12) | 8 (14) | 4 (4) | 5 (6) | 4 (5) | 12 (19)
Bone infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 13 (13) | 13 (14) | 8 (9) | 6 (7) | 2 (2) | 3 (3) | 4 (5)
Catheter related infection (Infections and infestations) | 8 (9) | 29 (32) | 37 (45) | 26 (29) | 21 (27) | 14 (19) | 13 (17) | 34 (40)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (5)
Encephalitis infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalomyelitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Endocarditis infective (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 12 (12) | 34 (38) | 31 (39) | 14 (15) | 17 (20) | 7 (7) | 14 (17) | 49 (63)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 2 (2) | 6 (7) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Gum infection (Infections and infestations) | 0 (0) | 8 (8) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 7 (8)
Hepatic infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 227 (312) | 489 (962) | 463 (906) | 249 (467) | 298 (643) | 134 (298) | 142 (341) | 434 (1120)
Infective myositis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Joint infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Lung infection (Infections and infestations) | 4 (4) | 74 (91) | 89 (103) | 53 (63) | 53 (59) | 28 (37) | 18 (19) | 73 (92)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (5)
Mucosal infection (Infections and infestations) | 1 (1) | 5 (5) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 41 (50) | 48 (53) | 22 (27) | 25 (27) | 6 (7) | 14 (16) | 44 (52)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Penile infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 14 (14) | 6 (7) | 9 (9) | 2 (4) | 1 (1) | 4 (5) | 4 (4)
Pleural infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 4 (5) | 7 (7) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 11 (11)
Sinusitis (Infections and infestations) | 0 (0) | 44 (51) | 38 (46) | 19 (26) | 26 (29) | 5 (8) | 8 (8) | 20 (22)
Skin infection (Infections and infestations) | 8 (9) | 32 (36) | 37 (40) | 22 (24) | 28 (33) | 7 (7) | 7 (8) | 37 (43)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Soft tissue infection (Infections and infestations) | 2 (2) | 5 (6) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Splenic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 5 (5) | 82 (107) | 94 (118) | 59 (69) | 61 (83) | 17 (24) | 15 (18) | 86 (107)
Urethral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (6) | 31 (34) | 19 (24) | 22 (30) | 17 (21) | 8 (8) | 8 (11) | 26 (31)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vulval infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 14 (14) | 6 (6) | 5 (6) | 9 (10) | 3 (3) | 2 (2) | 11 (11)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraoperative ocular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraoperative respiratory injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 8 (8) | 7 (9) | 9 (13) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 7 (7)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 17 (17) | 23 (24) | 6 (6) | 9 (12) | 8 (9) | 5 (5) | 2 (4) | 23 (31)
Alanine aminotransferase increased (Investigations) | 174 (177) | 453 (1316) | 443 (1235) | 207 (500) | 250 (689) | 123 (362) | 107 (372) | 310 (1009)
Alkaline phosphatase increased (Investigations) | 0 (0) | 5 (6) | 9 (10) | 11 (12) | 3 (3) | 1 (1) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 59 (60) | 220 (335) | 188 (278) | 89 (133) | 91 (137) | 54 (82) | 58 (98) | 164 (288)
Blood bilirubin increased (Investigations) | 20 (20) | 77 (90) | 53 (89) | 28 (42) | 30 (42) | 26 (34) | 16 (19) | 43 (52)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 7 (7) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 50 (50) | 41 (58) | 40 (48) | 31 (35) | 24 (28) | 17 (23) | 12 (17) | 29 (36)
GGT increased (Investigations) | 28 (29) | 49 (79) | 21 (22) | 10 (13) | 17 (26) | 10 (13) | 12 (17) | 27 (45)
INR increased (Investigations) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Investigations - Other, specify (Investigations) | 4 (4) | 8 (10) | 9 (11) | 12 (15) | 6 (9) | 3 (3) | 0 (0) | 12 (17)
Lipase increased (Investigations) | 28 (29) | 38 (43) | 7 (10) | 8 (9) | 10 (15) | 5 (5) | 14 (17) | 28 (42)
Lymphocyte count decreased (Investigations) | 8 (9) | 56 (94) | 72 (117) | 24 (39) | 43 (95) | 14 (24) | 23 (50) | 46 (118)
Neutrophil count decreased (Investigations) | 166 (172) | 708 (2226) | 727 (2182) | 375 (1101) | 429 (1457) | 184 (620) | 201 (731) | 570 (2396)
Platelet count decreased (Investigations) | 108 (111) | 262 (405) | 199 (297) | 108 (143) | 151 (236) | 62 (89) | 79 (142) | 274 (567)
Serum amylase increased (Investigations) | 17 (17) | 17 (19) | 6 (7) | 5 (5) | 7 (11) | 4 (4) | 4 (5) | 20 (24)
Weight gain (Investigations) | 9 (9) | 17 (18) | 16 (18) | 10 (12) | 5 (7) | 5 (5) | 3 (3) | 20 (22)
Weight loss (Investigations) | 7 (7) | 11 (12) | 7 (8) | 6 (10) | 5 (5) | 4 (4) | 5 (5) | 16 (17)
White blood cell decreased (Investigations) | 106 (110) | 304 (765) | 345 (903) | 160 (354) | 188 (547) | 89 (235) | 113 (337) | 268 (927)
Acidosis (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 4 (4) | 2 (2) | 5 (6) | 2 (2) | 1 (1) | 6 (6)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 16 (16) | 42 (51) | 35 (51) | 23 (41) | 30 (37) | 7 (8) | 22 (26) | 67 (91)
Dehydration (Metabolism and nutrition disorders) | 19 (19) | 54 (67) | 51 (62) | 33 (38) | 45 (55) | 16 (17) | 21 (26) | 83 (105)
Glucose intolerance (Metabolism and nutrition disorders) | 7 (7) | 4 (5) | 3 (4) | 2 (2) | 6 (6) | 3 (6) | 0 (0) | 9 (13)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 77 (77) | 52 (57) | 45 (50) | 44 (52) | 37 (44) | 21 (27) | 18 (21) | 71 (102)
Hyperkalemia (Metabolism and nutrition disorders) | 22 (22) | 19 (19) | 17 (19) | 5 (5) | 13 (15) | 4 (4) | 4 (4) | 25 (26)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 7 (7) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 (8) | 8 (9) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 3 (3) | 7 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 (26) | 66 (75) | 34 (37) | 17 (17) | 13 (15) | 10 (10) | 12 (12) | 41 (52)
Hypocalcemia (Metabolism and nutrition disorders) | 38 (38) | 35 (36) | 34 (35) | 25 (25) | 14 (15) | 11 (11) | 13 (14) | 38 (40)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 61 (73) | 16 (19) | 17 (21) | 7 (8) | 13 (16) | 10 (10) | 40 (47)
Hypokalemia (Metabolism and nutrition disorders) | 70 (70) | 107 (127) | 115 (135) | 53 (70) | 64 (80) | 35 (49) | 30 (40) | 138 (191)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 77 (78) | 75 (90) | 62 (68) | 41 (43) | 42 (47) | 19 (20) | 18 (20) | 66 (80)
Hypophosphatemia (Metabolism and nutrition disorders) | 20 (20) | 13 (13) | 21 (21) | 12 (12) | 7 (7) | 4 (4) | 4 (4) | 20 (20)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 14 (14) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (11) | 3 (3) | 2 (5) | 3 (4) | 1 (1) | 1 (2) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (12) | 12 (12) | 15 (17) | 6 (6) | 2 (2) | 5 (6) | 18 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (11) | 6 (6) | 1 (3) | 8 (8) | 4 (4) | 3 (3) | 8 (8)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 16 (16) | 9 (10) | 7 (7) | 5 (6) | 7 (7) | 2 (3) | 2 (3) | 12 (12)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (14) | 34 (38) | 22 (25) | 14 (16) | 18 (25) | 4 (5) | 4 (5) | 24 (32)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arachnoiditis (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 5 (5) | 6 (7) | 7 (7) | 1 (1) | 6 (6) | 2 (2) | 1 (1) | 16 (19)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (10) | 16 (19) | 21 (24) | 11 (17) | 23 (26) | 6 (6) | 4 (7) | 19 (30)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
IVth nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Ischemia cerebrovascular (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 8 (8) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 10 (10)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 4 (8) | 1 (1) | 2 (2) | 4 (5)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 38 (38) | 68 (105) | 52 (89) | 43 (76) | 39 (64) | 27 (46) | 22 (41) | 79 (141)
Peripheral sensory neuropathy (Nervous system disorders) | 29 (29) | 57 (94) | 41 (78) | 20 (42) | 38 (56) | 21 (29) | 9 (14) | 54 (85)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 12 (12) | 9 (9) | 11 (12) | 5 (5) | 13 (16) | 4 (5) | 7 (7) | 20 (24)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 3 (4)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 7 (7) | 8 (11) | 10 (10) | 6 (6) | 6 (6) | 0 (0) | 2 (2) | 8 (8)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (4) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 3 (3) | 2 (5)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 3 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 0 (0) | 6 (10) | 8 (11) | 4 (4) | 5 (7) | 1 (1) | 3 (3) | 6 (7)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 2 (2) | 10 (11) | 5 (8) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 4 (4) | 6 (9) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 4 (4)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (9) | 2 (2) | 0 (0) | 2 (2) | 1 (4) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (11) | 9 (12) | 5 (7) | 5 (5) | 6 (7) | 3 (4) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 13 (13) | 16 (16) | 10 (14) | 10 (11) | 2 (2) | 2 (2) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 5 (5) | 5 (7) | 5 (7) | 1 (1) | 3 (3) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 3 (4) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 9 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 30 (32) | 25 (26) | 11 (14) | 14 (14) | 9 (14) | 10 (10) | 28 (34)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 13 (13) | 4 (4) | 4 (4) | 5 (5) | 0 (0) | 4 (5) | 9 (9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 21 (23) | 20 (21) | 7 (8) | 10 (10) | 4 (6) | 5 (6) | 22 (24)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8) | 15 (16) | 8 (8) | 1 (1) | 2 (2) | 0 (0) | 11 (12)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (11) | 7 (9) | 4 (4) | 12 (13) | 3 (3) | 5 (6) | 15 (18)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (12) | 4 (4) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 10 (12)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 5 (5)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 30 (31) | 18 (18) | 29 (31) | 8 (8) | 13 (15) | 6 (12) | 5 (6) | 30 (35)
Hypotension (Vascular disorders) | 10 (10) | 17 (18) | 10 (10) | 7 (7) | 8 (8) | 2 (2) | 1 (1) | 18 (21)
Thromboembolic event (Vascular disorders) | 17 (17) | 9 (9) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 5 (6)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 6 (6) | 3 (4) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 3 (3)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.